CLINICAL TRIAL: NCT06550271
Title: The Bioavailability of Compounded and Generic Rapamycin in Normative Aging Individuals: A Retrospective Study and Review With Clinical Implications
Brief Title: The Bioavailability of Compounded and Generic Rapamycin in Normative Aging Individuals
Status: Completed | Type: Observational
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Other Study IDs: ALRx005
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Aging
Keywords: Bioavailability; Rapamycin; Aging; Longevity; Sirolimus; Healthy aging; age-related conditions; energy improvement
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compounded Rapamycin: Participants in this group were receiving Compounded Rapamycin (dosages include 5, 10, or 15mg) once per week
  Interventions: Drug: Rapamycin
- Generic Rapamycin: Participants in this group were receiving Generia Rapamycin (dosages include 2,3,6, or 8mg) once per week
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Rapamycin in 2 different dosage forms (compounded and generic)
  Other Names: Sirolimus; Rapamune; Rapacan; Siromus; Raparen; Rapasim; Sirova

SUMMARY:
This study collected real-world evidence to better understand and define the relative bioavailability ratio between compounded rapamycin and generic rapamycin, with a specific focus on relative efficacy in increasing rapamycin levels in the blood (blood rapamycin levels).

ELIGIBILITY:
Inclusion Criteria:

* Receive AgelessRx's standard Rapamycin treatment protocol
* Opted to complete at least 1 blood draw at their local Quest Lab

Exclusion Criteria:

* Not approved for current AgelessRx standard Rapamycin treatment
* History of uncontrolled disease
* Unable to complete at least 1 blood draw at their local Quest Lab

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who sought rapamycin prescription for longevity support, pain reduction, energy improvement, weight loss, mood improvement, sleep improvement, or oral health improvement were included in the study. To be eligible to receive AgelessRx's standard rapamycin treatment protocol, participants had to be ≥40 years of age, without a history of uncontrolled disease. All patients treated with rapamycin and opted for at least one blood draw test between May 1, 2023, and December 15, 2023, were included in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
define the relative bioavailability ratio between compounded rapamycin and generic rapamycin | 8 months
  define the relative bioavailability ratio between compounded rapamycin and generic rapamycin, with a specific focus on relative efficacy in increasing rapamycin levels in the blood (blood rapamycin levels).

CONTACTS AND LOCATIONS:
Overall Officials: Sajad Zalzala, MD, Study Director — AgelessRx
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided